CLINICAL TRIAL: NCT05558592
Title: Evaluation of the Effects of Orange Consumption on Carbohydrate and Lipid Metabolism in Subjects With MAFLD (Metabolic Associated Fatty Liver Disease)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Cisternino Anna Maria (Unknown); Valeria Tutino (Unknown); Valentina De Nunzio (Unknown); Roberta Rinaldi (Unknown)
Responsible Party: Principal Investigator, Maria Notarnicola, principal investigator, biologist, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC2022_prg.15
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Disease; Fatty Liver, Nonalcoholic
MeSH Terms: conditions — Metabolic Diseases; Non-alcoholic Fatty Liver Disease | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment_group (Experimental)
  Interventions: Dietary Supplement: Dietary supplementation with fresh oranges
- Control_group (Active Comparator)
  Interventions: Dietary Supplement: Balanced Diet without oranges

INTERVENTIONS:
Dietary Supplement: Dietary supplementation with fresh oranges — the subjects enrolled in this group, will have to consume 400gr of oranges "Navelina" net of waste / day / per person for a month. The oranges will be provided, to each participant, by the IRCCS "Saverio de Bellis".
  Arms: Treatment_group
Dietary Supplement: Balanced Diet without oranges — the subjects enrolled in this group, will have to consume 400 gr of fruit (with the exception of citrus fruits) net of waste / day / per person for a month.
  Arms: Control_group

SUMMARY:
Given the current increase in the incidence of dyslipidemia and obesity in the general population, there is a strong interest in identifying dietary factors capable of preventing the onset of metabolic diseases or at least capable of reducing metabolic risk. Several experimental evidences have shown that improving the carbohydrate and lipid profile in subjects at risk can reduce mortality linked to cardiovascular, neurodegenerative diseases and cancer. The diet is, therefore, an effective prevention tool in combating diseases related to metabolism, such as MAFLD (Metabolic Associated Fatty Liver Disease). In particular, fruit with its high content of polyphenols has been shown to exert a high anti-inflammatory, antithrombotic and antiproliferative action.

Polyphenols extracted from oranges of the "Tacle" variety have demonstrated in vitro an inhibitory action of cholesterol synthesis. In addition, the consumption of orange juice has been shown to improve the serum lipid profile of obese subjects, as well as "hesperedine", a flavonoid mainly present in oranges is able to reduce the proliferative activity of MCF-7 (human breast cancer cell line with estrogen, progesterone and glucocorticoid receptors) cells.

ELIGIBILITY:
Inclusion Criteria:

* age > 30 years and <65 years
* diagnosis of MAFLD on the basis of clinical and instrumental parameters

Exclusion Criteria:

* gastroesophageal reflux diseases;
* inflammatory bowel diseases; oncological diseases;
* serious medical conditions that may impair participation in the trial;
* people who follow a special diet or who use anticoagulants;
* subjects unable to follow a diet for religious or other reasons.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
variation in lipidomic profile | 1 year
  change in membrane lipidomic profile and
changes in MAFLD score | 1 year
  changes in MAFLD score at the end of the treatment period from baseline - this score is evaluated as change in grade of steatosis Measurement of steatosis: The Controlled Attenuation Parameter (CAP) measurement was performed by a vibration-controlled elastography (VCTE) implemented on FibroScan® (Echosens, Paris, France). The CAP score is measured in decibels per meter (dB/m). Values < 215 dB/m corresponded to the absence of NAFLD; values between 215 and 250 dB/m indicated a mild NAFLD; values between 251 and 299 dB/m indicated a moderate NAFLD, while values ≥ 300 dB/m corresponded to a severe NAFLD.

SECONDARY OUTCOMES:
variation in antioxidant status | 1 year
  evaluation of antioxidant status and improvement of inflammatory parameters in order to reduce metabolic risk in subjects with MAFLD
changes in inflammatory parameters | 1 year
  and improvement of inflammatory parameters in order to reduce metabolic risk in subjects with MAFLD

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Saverio de Bellis, Castellana Grotte, BARI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ammollo CT, Semeraro F, Milella RA, Antonacci D, Semeraro N, Colucci M. Grape intake reduces thrombin generation and enhances plasma fibrinolysis. Potential role of circulating procoagulant microparticles. J Nutr Biochem. 2017 Dec;50:66-73. doi: 10.1016/j.jnutbio.2017.08.012. Epub 2017 Sep 1. PMID 29040837
- [Result] Tutino V, Gigante I, Milella RA, De Nunzio V, Flamini R, De Rosso M, Scavo MP, Depalo N, Fanizza E, Caruso MG, Notarnicola M. Flavonoid and Non-Flavonoid Compounds of Autumn Royal and Egnatia Grape Skin Extracts Affect Membrane PUFA's Profile and Cell Morphology in Human Colon Cancer Cell Lines. Molecules. 2020 Jul 23;25(15):3352. doi: 10.3390/molecules25153352. PMID 32718061
- [Result] Tutino V, De Nunzio V, Milella RA, Gasparro M, Cisternino AM, Gigante I, Lanzilotta E, Iacovazzi PA, Lippolis A, Lippolis T, Caruso MG, Notarnicola M. Impact of Fresh Table Grape Intake on Circulating microRNAs Levels in Healthy Subjects: A Significant Modulation of Gastrointestinal Cancer-Related Pathways. Mol Nutr Food Res. 2021 Nov;65(21):e2100428. doi: 10.1002/mnfr.202100428. Epub 2021 Sep 21. PMID 34495579
- [Result] Simpson EJ, Mendis B, Macdonald IA. Orange juice consumption and its effect on blood lipid profile and indices of the metabolic syndrome; a randomised, controlled trial in an at-risk population. Food Funct. 2016 Apr;7(4):1884-91. doi: 10.1039/c6fo00039h. PMID 26965492
- [Result] Akiyama S, Katsumata S, Suzuki K, Ishimi Y, Wu J, Uehara M. Dietary hesperidin exerts hypoglycemic and hypolipidemic effects in streptozotocin-induced marginal type 1 diabetic rats. J Clin Biochem Nutr. 2010 Jan;46(1):87-92. doi: 10.3164/jcbn.09-82. Epub 2009 Dec 29. PMID 20104270
- [Derived] Notarnicola M, Tutino V, De Nunzio V, Cisternino AM, Cofano M, Donghia R, Giannuzzi V, Zappimbulso M, Milella RA, Giannelli G, Fontana L. Daily Orange Consumption Reduces Hepatic Steatosis Prevalence in Patients with Metabolic Dysfunction-Associated Steatotic Liver Disease: Exploratory Outcomes of a Randomized Clinical Trial. Nutrients. 2024 Sep 20;16(18):3191. doi: 10.3390/nu16183191. PMID 39339791